CLINICAL TRIAL: NCT06712602
Title: Selective Glucocorticoid Receptor Antagonism in Alcohol Use Disorder: A Human Laboratory Study
Brief Title: PT150 Drug for Use in Alcohol Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pop Test Oncology LLC (Industry)
Collaborators: University of Kentucky (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 90580; R01AA030774 (NIH)
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Alcohol Use Disorder; Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; (11R,13S,17S)-11-(1,3-benzodioxol-5-yl)-17-hydroxy-13-methyl-17-prop-1-ynyl-1,2,6,7,8,11,12,14,15,16-decahydrocyclopenta(a)phenanthren-3-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PT150 with alcohol consumption then stress (Experimental): Following at least five days of maintenance on a randomized dose of PT150, participants will complete an experimental alcohol administration session. No less than 24 hours later, participants will then complete an experimental stress induction session.
  Interventions: Drug: alcohol; Behavioral: Stress-Induction; Drug: PT150
- PT150 with stress then alcohol consumption (Experimental): Following at least five days of maintenance on a randomized dose of PT150, participants will complete an experimental session involving stress induction. No less than 24 hours later, participants will then complete an experimental alcohol administration session.
  Interventions: Drug: alcohol; Behavioral: Stress-Induction; Drug: PT150

INTERVENTIONS:
Drug: alcohol — During the alcohol administration session participants will receive a single administration of alcohol (0.5 g/kg) mixed with lemon lime soda. Participants will consume the drink within 5 min.
Behavioral: Stress-Induction — The stress-induction procedure is the Cold Pressure Test [CPT]) stressor. The bilateral foot CPT requires participants to submerge both feet in ice-cold water (24°C) for 3 minutes.
Drug: PT150 — Participants will ingest PT150 (0, 225, 450 mg) twice daily (e.g., 0800, 2000h) for 5 five days prior to the conduct of the experimental sessions. The sequence of PT150 doses will be quasi-random such that participants will be maintained on the lower dose of PT150 (i.e., 225 mg twice/day) before the higher dose.

SUMMARY:
The goal of this study is to learn if PT150 can reduce the behavioral and physical effects of stress, alcohol, and alcohol use in people with alcohol use disorder.

DETAILED DESCRIPTION:
The Investigators will conduct behavioral testing in an individual room with a lounge chair and laptop computer for completing the questionnaires, along with supplies for the bilateral foot CPT. Computerized data collection increases the accuracy of data collection and efficiency of data management. Participants will remain seated in the lounge chair for the duration of the session. Procedures Specific to the Stress-Induction Session Stress-Induction. The stress-induction procedure is the Cold Pressure Test [CPT]) stressor. The bilateral foot CPT requires participants to submerge both feet in ice-cold water (2-4°C) for 3 minutes . The Investigators will inform participants the cold water, while painful, will not cause tissue damage. The Investigators will further instruct participants a same-sex research assistant and medical staff will monitor them for their safety. Participants will not know how much time remains in the procedure (i.e., no clocks, watches or electronic devices allowed). The Investigators will record behavioral (i.e., alcohol demand, craving, mood, and subjective effects) and neuroendocrinological (i.e., salivary cortisol) responses as noted in Table 2. Stress-induction procedures are safe, and reliably elicit behavioral and neuroendocrinological responses in controls and patients with AUD, including those with PTSD. The Investigators will demonstrate the internal validity of the stress-induction procedure using a single visual analog scale anchored with adjective modifiers (0=Not at All to 100=Extremely): How STRESSED are you right now? Alcohol Demand. The Investigators will use a purchasing task to measure alcohol demand. Participants will report hypothetical consumption of their preferred alcohol beverage across a range of prices given they can only get the drinks from a single source and would have to consume all of them in a single sitting. Single doses of their preferred alcohol beverage will be available across 14 prices (i.e., $0.00 [Free], $0.01 $0.03, $0.30, $1, $3, $10, $30, $100, $300, $1,000). All choices will be hypothetical, and the Investigators will not administer any alcohol during this task. Alcohol purchasing tasks are sensitive to stress manipulations. Craving and Mood Questionnaires. The Investigators will use two instruments to assess craving. First, the Investigators will use the Alcohol Urge Questionnaire. Second, the Investigators use a set of four unidimensional visual analog scales: 1) How strong is your craving to drink alcohol? 2) If I could drink alcohol now, I would drink it; 3) It would be hard to turn down a drink right now; and 4) Having a drink would make things just perfect. The Investigators will use the short form of the Profile of Mood States. The POMS-SF uses five-point scales (Not at All to Extremely) to measure six aspects of mood (Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment). The Alcohol Urge Questionnaire and POMS-SF are sensitive to stress manipulations. Salivary Cortisol. The Investigators will collect salivary cortisol samples before and periodically after the stress-induction procedure for 120 minutes using cotton swab Salivettes®. The Investigators will store the samples at room temperature until the end of the experimental session and then at -80°C until analyzed using the standard University of Kentucky laboratory assessment. Safety Measures. The Investigators will record heart rate and blood pressure before the stress-induction procedure and afterwards for 120 mins. Procedures Specific to the Alcohol Administration Session Alcohol Challenge. During this session, participants will receive a single administration of alcohol (0.5 g/kg) mixed with lemon lime soda. The Investigators will instruct participants to consume the drink within 5 min. The Investigators will assess the behavioral and physiological effects before alcohol administration (Baseline) and afterwards for 120 mins using the measures described below (Table 2). The Investigators selected this dose because, in our experience, it is behaviorally active, well tolerated, and raises breath alcohol concentration ([BAC] for approximately 2.5-3.0 hours. Alcohol Demand. The Investigators will use the purchasing task described above but modify it to reflect the hypothetical choices between the drink they sampled across varying prices. The Investigators have shown hypothetical alcohol choices are an orderly function of price and are sensitive to Section 9 Page 5 of 15 90580 putative pharmacotherapies. Craving, Mood, and Subjective-Effect Questionnaires. The Investigators will use four standardized subjective-effects questionnaires to measure various aspects of mood and alcohol effects: 1) Biphasic Alcohol Effects Scale; 2) Subjective High Assessment Scale; 3) Alcohol Urge Questionnaire; and 4) of Mood States Short Form. The Investigators will use the set of 4 unidimensional visual analog scales described above. The Investigators will also use a locally developed 10-item Drug Effect Questionnaire. Participants rate each item using visual analog scales anchored with adjective modifiers (0=Not at All to 100=Extremely) to rate the effects of the drink: Any Effects, Bad Effects, Drunk, Good Effects, Like Effects, Performance Impaired, Performance Improved, Stimulated, Talkative-Friendly, and Willing to Take Again. Performance Measure. The Investigators will assess motor coordination using a grooved pegboard task (Lafayette Instruments, Lafayette, IN). During this task, participants place pegs into keyhole-shaped holes. The grooved pegboard contains a rectangular metal surface with 25 holes arranged in five rows of five holes. Each of the holes has a rounded side and smaller square side (a groove). The orientation of the groove in each hole varies so that no two adjacent holes have the same orientation. Each peg is 3 mm in diameter and 2.5 cm long and has a rounded side and grooved side. Pegs fit into the holes like a key would fit into a lock. Participants are required to pick up pegs one at a time and place them in holes. They fill one row at a time and work from left to right. A trial on the grooved pegboard task was completed when all 25 holes were filled, and the time to complete a trial was the measure of interest. A grooved pegboard test consisted of four trials, and the time to complete each of the trials was averaged to calculate the measure of motor coordination. The grooved pegboard task is sensitive to the effects of. Salivary Cortisol. The Investigators will collect salivary cortisol samples before and periodically after alcohol administration as shown in Table 2. Safety Measures. The Investigators will record heart rate, blood pressure, and BAC levels before administering the ALC dose and afterwards for 120 mins. Procedures Specific to Assessing Alcohol Use, Craving, and Stress in the Natural Ecology Participants will access a REDCap survey daily to report the number of drinks consumed in the past day and to complete the Alcohol Urge Questionnaire, POMS-SF, Perceived Stress Questionnaire, and the single-item sleep quality questionnaire. The Investigators will also use the REDCap survey to monitor adverse events. The Investigators will calculate the number of heavy drinking days for each participant (males = 5 standard drinks, females =4 standard drinks; NIAAA, 2017). The Investigators have used similar procedures in the past to measure the effects of putative pharmacotherapies for AUD in the natural environment. Follow-Up Visit and Discharge from Study, the Investigators will schedule participants for a follow-up visit approximately one week after the last experimental session (i.e., those completing the study) or the final session completed (i.e., those not completing the study; Table 1). During this visit the Investigators will gather much of the same information recorded during the Pre-Participation Screening (e.g., drug-use questionnaire, heart rate and blood pressure, urine drug test). The Investigators will also query participants regarding how they used payments dispersed after their final experimental session. Participants will complete the Perceived Research Burden Assessment and Coercion Assessment Scale during the follow-up visit to measure their overall study experience. Data Analysis, the Investigators will analyze data as raw scores unless noted otherwise. The Investigators will replace participants who do not complete the study until the Investigators accrue 34 completers to ensure sufficient statistical power. Statistical significance refers to p equal to or less than 0.05. The Investigators predict: 1) stress induction will increase cortisol, alcohol demand and negative mood, and PT150 will attenuate these responses, 2) alcohol will increase alcohol demand and produce prototypical subjective effects and PT150 will attenuate these effects, and 3) PT150 will decrease drinking, craving, and stress in the natural ecology. Exploratory analyses will determine if: 1) responses/changes differ in females and males; 2) baseline cortisol or stress levels predict behavioral or neuroendocrinological responses to stress and attenuation by PT150; and 3) behavioral and neuroendocrinological responses and attenuation by PT150 during the stress-induction session predict changes in the natural ecology. Stress-Induction Session (Specific Aim 1). The Investigators will analyze data from the purchase task (i.e., alcohol demand) using derived and curve-observed measures. Derived measures include demand intensity (Q0; consumption at unconstrained price) and demand elasticity (a measure of sensitivity of consumption to changes in price) and will be computed using the exponential demand equation LogQ=Log Q0+k(e^(-a Q0C)-1. The independent variable C is cost (price/dose), the dependent variable Q is consumption (doses purchased at a particular price), and the scaling parameter k indicates the range of LogQ in the observed data. Free parameters are Q0 (demand intensity) and a (demand elasticity). Should the Investigators observe zero-dense data, the Investigators will consider using a modified exponentiated form of the demand equation. Outcome measures include Pmax (price at maximum consumption), Omax (maximum consumption) and breakpoint (Breakpoint-1; the price of last non-zero demand), Q0 (demand intensity) and a (demand elasticity). Behavioral (e.g., alcohol demand, craving, mood, and subjective effects) and neuroendocrinological (e.g., salivary cortisol) outcomes from the stress-induction session will be analyzed with generalized linear mixed models (GLMM), allowing us to statistically account for the longitudinal nature of the data. GLMM are virtually identical to repeated measures ANOVA when no data are missing but can appropriately handle non-normal outcomes and allow the specification of numerous covariance structures. The Investigators will enter PT150 dose (0, 450, 900 mg), Time (Baseline, 0, 10, 20, 30, 45, 60, 90, 120) minutes after stress-induction or alcohol administration), and their interaction into the models as predictors. The Investigators will use severity of AUD (moderate, severe) and baseline Section 9 Page 6 of 15 90580 measures of quantity and frequency (e.g., drinks/drinking day, drinking days/month) as a time-invariant predictor in all models to control for levels of alcohol use. The Investigators will use design matrix for testing custom hypotheses regarding the outcome response profiles over time (e.g., linear, quadratic, or piecewise change) and whether these trajectories differ by PT150 dose to infer a significant attenuation of the effects of stress-induced responses if the main effect of PT150 or the interaction of PT150 and Time attains statistical significance. If the interaction of PT150 and Time attains statistical significance, the Investigators will use Tukey's HSD corrected for multiple comparisons to determine the locus of the effect by making appropriate pair-wise comparisons. The Investigators will also calculate area-under-the curve (AUC) using the trapezoidal method for appropriate measures (e.g., cortisol) and analyze these data similarly excluding Time from the model (Scheff et al., 2011). Alcohol Challenge Session (Specific Aim 2). The Investigators will analyze data (alcohol demand, craving, subjective effects, breath-alcohol) from the ALC challenge session as described above. Alcohol Use, Craving and Stress in the Natural Ecology (Specific Aim 3). The Investigators will analyze alcohol use in the natural ecology as total number of drinks and heavy drinking days during each maintenance phase. The Investigators will average data from the Alcohol Urge Questionnaire, POMS-SF, single-item sleep quality questionnaire, and Perceived Stress Questionnaire across maintenance days on each PT150 dose. The Investigators will analyze these data with GLMM with PT150 (0, 450, 900 mg/day) as the sole within-subject factor. The Investigators will infer a significant increase or decrease if the main effect of the PT150 attains statistical significance. If the omnibus test is significant, the Investigators will use Tukey's HSD corrected for multiple comparisons to make comparisons between means. Exploratory Analysis (Exploratory Aims). The Investigators will use multivariate latent curve models to concurrently model the same longitudinal outcomes collected following stress-induction and the alcohol sample dose to compare the growth processes (i.e., intercept, slope) of these outcomes. Sex is the primary biological variable of interest because the effects of selective GR antagonists differed in males and females in preclinical. Safety and Adverse Events. The Investigators will use GLMM with PT150 group (0, 450, 900 mg/day) and Time (Pre- versus Post-Participation). The Investigators will infer significant changes if the main effects of PT150 group or Time, as well as the interaction of these variables, attain statistical significance. If the interaction of PT150 and Time attains statistical significance, the Investigators will use Tukey's HSD corrected for multiple comparisons with the mean square error term to make appropriate pair-wise comparisons. The Investigators will record adverse event frequency during maintenance as a count variable (i.e., number of side effects reported). Comparison by dose condition will use GLMM with a log link (i.e., Poisson distribution) and dose as a time-varying covariate. Power and Sample Size. The Investigators used the results of a previous human laboratory study in participants with AUD to estimate an appropriate sample size for detecting an effect of GR antagonism on experimentally induced increases in craving. Mifepristone reduced experimentally induced increases in alcohol craving (mean Cohen's f = 0.32). The Investigators used the results of a meta-analysis of human laboratory studies of alcohol self-administration and craving to determine an appropriate sample size for the proposed study to detect whether PT150 attenuates the acute pharmacodynamic effects of alcohol. Naltrexone decreased alcohol consumption and self-reported craving relative to placebo with an average estimated effect size of Hedges' g=-0.28. The previous study described above with mifepristone reported reductions in drinking in the natural ecology with an average estimated effect size of Cohen's f = 0.26. Considering the crossover design and 3 levels of PT150 (0, 450, 900 mg/day), enrolling 34 participants will provide power >0.85 (alpha=0.05, nQuery®) for us to detect an effect of PT150 on experimentally-induced stress responses (Specific Aim 1), the pharmacodynamic effects of alcohol (Specific Aim 2), and alcohol use in the natural ecology (Specific Aim 3) with an effect size similar to those observed previously (Cohen's f=0.25, power=0.80, alpha=0.05, nQuery®). The proposed statistical procedures (i.e., GLMM) can also accommodate missing data via maximum and quasi-likelihood estimation algorithms. The Investigators will include data available from participants who do not complete to further ensure adequate statistical power to detect the effects of PT150 on the primary outcomes. Enrolling 34 participants (17 females, 17 males) is also sufficient to determine whether the effects of PT150 differ as a function of sex. A preclinical study determined the effects of a range of doses of CORT113176, a selective GR antagonist, on alcohol self-administration in male and female (9-10/sex) rats and found a significant effect of sex. Finally, enrolling 34 participants is also sufficient to determine if baseline cortisol or stress levels predict behavioral or neuroendocrinological responses to stress and attenuation by PT150; and whether the behavioral and neuroendocrinological responses and attenuation by PT150 during the stress-induction session predict changes drink in the natural ecology (Exploratory Aims). One of the studies described above reported reductions in experimentally induced alcohol craving observed with mifepristone in the laboratory predicted reductions in the number of drinks per drinking day in the natural ecology (R2=0.11, p=0.017, Cohen's f=0.352).

ELIGIBILITY:
Inclusion Criteria:

Meet diagnostic criteria for AUD (moderate or severe) per the Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-5)

Not seeking treatment at the time of the study

English-speaking

Between the ages of 21 and 55 years (individuals under 21 are excluded based on the recommendations of NIAAA that alcohol should not be administered to individuals under the legal drinking age)

Abstinent from alcohol no more than 3 days per week on average

Physically and psychiatrically healthy other than the diagnoses for AUD or tobacco use disorder

ECG, read by cardiologist, within normal limits

Body mass index of 19 - 35

Using an effective form of birth control (e.g., birth control pills, surgical sterilization, condoms, IUD, cervical cap with a spermicide or abstinence) if female

Able to abstain from ALC for 12 hours prior to sessions

No contraindications to ALC or PT150

Exclusion Criteria:

Meet diagnostic criteria for SUDs, save nicotine, other than AUD that in the opinion of a study physician would require medical intervention (e.g., opioid use disorder) or compromise the well-being of the participant

Have abnormal blood chemistry, complete blood count or urinalysis values deemed clinically significant

Have a history of serious physical disease or current physical disease (e.g., impaired cardiovascular functioning, histories of seizure, head trauma or CNS tumors)

Have a current or past history of psychiatric disorder that would interfere with participation (e.g., psychotic [schizophrenia, schizoaffective]), bipolar, major depressive disorder)

Have had suicidal ideations in the past 90 days

Pregnant or nursing

Are unwilling/unable to comply with study procedures

Participants scoring >6 on the Clinical Institute Withdrawal Assessment for Alcohol Revised (CIWA-Ar); the CIWA-Ar will be administered prior to each experimental session participants who score >6 will be excluded further participation.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in salivary cortisol (alcohol) | Baseline, week 1, week 2, week 3, and follow up (up to 34 days)
  Salivatory samples will be collected before and periodically after the alcohol challenge procedure for 120 minutes using cotton swab salivettes.
Change in salivary cortisol (stress induction) | Baseline, week 1, week 2, week 3, and follow up visit (up to 34 days)
  Salivatory samples will be collected before and periodically after the stress induction procedure for 120 minutes using cotton swab salivettes.
Change in Alcohol Demand (stress induction) | Baseline, and sessions 1 - 3 (up to 30 days)
  A drug purchasing task will be used to determine how many hypothetical doses of their preferred alcohol beverage participants would purchase across varying prices.
Change in Alcohol Demand (alcohol) | Baseline, and sessions 1 - 3 (up to 30 days)
  A drug purchasing task will be used to determine how many hypothetical doses of the alcoholic beverage given during the session participants would purchase across varying prices.
Change in Mood (Alcohol) | Baseline, and sessions 1 - 3 (up to 30 days)
  The short form of the Profile of Mood States. The POMS-SF uses five-point scales (Not at All to Extremely) to measure six aspects of mood (Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment).

SECONDARY OUTCOMES:
Change in Heart Rate (Stress) | Baseline, sessions 1 - 3, and follow up visit (up to 34 days)
Change in Heart Rate (Alcohol) | Baseline, sessions 1 - 3, and follow up visit (up to 34 days)
Change in blood pressure (stress) | Baseline, sessions 1 - 3, and follow up visit (up to 34 days)
Change in blood pressure (alcohol) | Baseline, sessions 1 - 3, and follow up visit (up to 34 days)
Change in motor coordination | Baseline, and sessions 1 - 3 (up to 30 days)]
  Motor coordination will be measured using a grooved pegboard task during the alcohol intervention. Participants place pegs into keyhole-shaped holes. Participants are required to pick up pegs one at a time and place them in holes. time to complete a trial will be measured. The test consists of four trials, and the time to complete each of the trials will be averaged to calculate the measure of motor coordination.
Change in blood alcohol concentration | Baseline, and sessions 1 - 3 (up to 30 days)
  Blood alcohol levels will be measured before and after administration of the alcohol dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fillmore, PhD, Principal Investigator — Uiversity of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No